CLINICAL TRIAL: NCT04945564
Title: Covid-19 Patients Management During Home Isolation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, A. Sedky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/036-2021
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Oxygen; Physical Therapy Modalities; Oxygen Inhalation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen therapy and physical therapy (Experimental)
  Interventions: Procedure: Oxygen therapy and physical therapy
- Oxygen therapy (Active Comparator)
  Interventions: Device: Oxygen therapy

INTERVENTIONS:
Procedure: Oxygen therapy and physical therapy — Patients receive oxygen therapy and physical therapy
  Arms: Oxygen therapy and physical therapy
Device: Oxygen therapy — Patients receive oxygen therapy
  Arms: Oxygen therapy

SUMMARY:
The study will investigate management of Covid-19 patients in home isolation.

DETAILED DESCRIPTION:
A clinical trial concerned with the treatment of home isolated COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 patients American Society of Anesthesiologists (ASA) class I >= 21 years old <= 40 years old

Exclusion Criteria:

* Not being consistent with home-isolation regimen

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Time for recovery of pH | 24 hours
  Acidity Potential Hydrogen
Time for recovery of PaO2 | 24 hours
  Partial Pressure of Oxygen
Time for recovery of PaCO2 | 24 hours
  Partial Pressure of Carbon Dioxide
Chest CT scan | Baseline
  Chest computed tomography scan
Chest CT scan | 1 day post-treatment
  Chest computed tomography scan

SECONDARY OUTCOMES:
Time for recovery of Temperature | 24 hours
  vital sign
Time for recovery of Respiratory Rate | 24 hours
  vital sign
Time for recovery of Oxygen Saturation | 24 hours
  vital sign
Time for recovery of Heart Rate | 24 hours
  vital sign
Time for recovery of Blood Pressure | 24 hours
  vital sign

CONTACTS AND LOCATIONS:
Locations (1):
- A. Sedky, Cairo, Egypt